CLINICAL TRIAL: NCT05175144
Title: Diagnostic Performance of "Emergency Department Assessment of Chest Pain Score" in Patients With Acute Chest Pain.
Brief Title: Diagnostic Performance of "Emergency Department Assessment of Chest Pain Score"
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Arwa Salah Abdelaziz Ali, resident, Assiut University
Other Study IDs: Chest Pain Score
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Acute Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate whether EDACS performed during triage to assess patients with chest pain could improve the predictive validity of triage for an acute cardiovascular event.

DETAILED DESCRIPTION:
Chest pain is common reasons for presentation to the emergency department (ED).Up to 6.3% of emergency department (ED) visits are related to chest pain. Causes of chest pain range from musculoskeletal chest pain to potentially life-threatening emergencies as acute coronary syndrome(ACS), aortic dissection or pulmonary embolism. Therefore, accurate and fast risk stratification is paramount in the acute management, mainly to identify those patients with immediate risk of complications, as those with an ACS. Those patients are challenging to discriminate, as there is a variety of clinical manifestations.

Chest pain is considered to be an acute chest pain, described as pain, pressure, tightness, or burning as outlined in the guidelines Chest pain equivalent symptoms may include dyspnea, left arm, and epigastric pain.

Triage helps recognize the urgency among patients. An accurate triage decision helps patients receive the emergency service in the most appropriate time. Various triage systems have been developed and verified to assist healthcare providers to make accurate triage decisions. Despite good levels of specificity, the available triage systems appear to have suboptimal sensitivities that cannot adequately prioritize patients with acute cardiovascular diseases. The Emergency Department Assessment of Chest Pain Score (EDACS), through a standardized assessment of the patient's history and presenting symptoms only, provides good levels of sensitivity in stratifying time dependent acute cardiovascular diseases. The good discriminatory ability of EDACS, combined with its easy clinical applicability, could be used to overcome some of the limitations of triage systems in assessing chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old who admitted to ED complaining of chest pain.
* Chest pain is considered to be an acute chest pain, described as pain, pressure, tightness, or burning as outlined in the guidelines.
* Chest pain equivalent symptoms may include dyspnea, epigastric pain, and pain in the left arm.

Exclusion Criteria:

* Patients unable to complete the EDACS
* Posttraumatic chest pain
* Patients who did not give consent to participate

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient fulfilling the inclusion criteria can participating in our study . .
Sampling Method: Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of EDACS for detection of acute cardiovascular events in emergency department. | baseline

SECONDARY OUTCOMES:
Baseline characteristics for patients with acute cardiovascular events. | baseline

REFERENCES:
- [Background] Niska R, Bhuiya F, Xu J. National Hospital Ambulatory Medical Care Survey: 2007 emergency department summary. Natl Health Stat Report. 2010 Aug 6;(26):1-31. PMID 20726217
- [Background] Bayon Fernandez J, Alegria Ezquerra E, Bosch Genover X, Cabades O'Callaghan A, Iglesias Garriz I, Jimenez Nacher JJ, Malpartida De Torres F, Sanz Romero G; Grupo de Trabajo ad hoc de la Seccion de Cardiopatia Isquemica y Unidades Coronarias de la Sociedad Espanola de Cardiologia. [Chest pain units. Organization and protocol for the diagnosis of acute coronary syndromes]. Rev Esp Cardiol. 2002 Feb;55(2):143-54. doi: 10.1016/s0300-8932(02)76574-3. Spanish. PMID 11852005
- [Background] Hinson JS, Martinez DA, Cabral S, George K, Whalen M, Hansoti B, Levin S. Triage Performance in Emergency Medicine: A Systematic Review. Ann Emerg Med. 2019 Jul;74(1):140-152. doi: 10.1016/j.annemergmed.2018.09.022. Epub 2018 Nov 22. PMID 30470513
- [Background] Zaboli A, Ausserhofer D, Sibilio S, Toccolini E, Bonora A, Giudiceandrea A, Rella E, Paulmichl R, Pfeifer N, Turcato G. Effect of the Emergency Department Assessment of Chest Pain Score on the Triage Performance in Patients With Chest Pain. Am J Cardiol. 2021 Dec 15;161:12-18. doi: 10.1016/j.amjcard.2021.08.058. Epub 2021 Oct 9. PMID 34635312
- [Background] Than M, Flaws D, Sanders S, Doust J, Glasziou P, Kline J, Aldous S, Troughton R, Reid C, Parsonage WA, Frampton C, Greenslade JH, Deely JM, Hess E, Sadiq AB, Singleton R, Shopland R, Vercoe L, Woolhouse-Williams M, Ardagh M, Bossuyt P, Bannister L, Cullen L. Development and validation of the Emergency Department Assessment of Chest pain Score and 2 h accelerated diagnostic protocol. Emerg Med Australas. 2014 Feb;26(1):34-44. doi: 10.1111/1742-6723.12164. Epub 2014 Jan 15. PMID 24428678
- [Background] Than MP, Pickering JW, Aldous SJ, Cullen L, Frampton CM, Peacock WF, Jaffe AS, Goodacre SW, Richards AM, Ardagh MW, Deely JM, Florkowski CM, George P, Hamilton GJ, Jardine DL, Troughton RW, van Wyk P, Young JM, Bannister L, Lord SJ. Effectiveness of EDACS Versus ADAPT Accelerated Diagnostic Pathways for Chest Pain: A Pragmatic Randomized Controlled Trial Embedded Within Practice. Ann Emerg Med. 2016 Jul;68(1):93-102.e1. doi: 10.1016/j.annemergmed.2016.01.001. PMID 26947800
- [Background] Flaws D, Than M, Scheuermeyer FX, Christenson J, Boychuk B, Greenslade JH, Aldous S, Hammett CJ, Parsonage WA, Deely JM, Pickering JW, Cullen L. External validation of the emergency department assessment of chest pain score accelerated diagnostic pathway (EDACS-ADP). Emerg Med J. 2016 Sep;33(9):618-25. doi: 10.1136/emermed-2015-205028. Epub 2016 Jul 12. PMID 27406833